CLINICAL TRIAL: NCT00117286
Title: An Open-Label, Multi-Center, Extension Study Investigating the Long-Term Safety and Tolerability of Degarelix One-Month Depots in Patients With Prostate Cancer
Brief Title: Extension Study Investigating the Long-Term Safety of Degarelix One-Month Depots in Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS14A
Record Dates: First submitted 2005-06-30; First posted 2005-07-06 (Estimated); Results first posted 2010-10-21 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2010-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Androgen ablation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Degarelix (60 mg to 160 mg) (Experimental): Participants who completed the CS14 study in the Degarelix 60 mg (20 mg/mL) arm continued that dose into the CS14A extension study. A protocol amendment in March 2006 changed the dosage to 160 mg (40 mg/mL) for all study participants.
  Interventions: Drug: Degarelix
- Degarelix (80 mg to 160 mg) (Experimental): Participants who completed the CS14 study in the Degarelix 80 mg (20 mg/mL) arm continued that dose into the CS14A extension study. A protocol amendment in March 2006 changed the dosage to 160 mg (40 mg/mL) for all study participants.
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — Drug supplied as a powder to be dissolved in the solvent for solution for injection. Degarelix given by subcutaneous injection every 28 days until the end of the study.
  Other Names: Degarelix acetate, FE200486

SUMMARY:
This was an extension study for the study FE200486 CS14 (NCT00116779). Each participant was to be treated until he was discontinued or withdrawn from the study, or a marketing authorization for degarelix had been obtained.

The study was terminated when all ongoing participants had been treated for at least 5 years.

DETAILED DESCRIPTION:
Participants who completed the main FE200486 CS14 study initially continued with the same dose in the FE200486 CS14A extension study. A protocol amendment changed the dosage to 160 mg (40 mg/mL) for all study participants.

The data include data from the participants who participated in both the main study (FE200486 CS14; NCT00116779) and the extension study FE200486 CS14A.

ELIGIBILITY:
Inclusion Criteria:

* Has given written consent prior to any study-related activity being performed. A study-related activity is defined as any procedure that would not have been performed during the normal management of the patient.
* Has completed study FE200486 CS14 through visit 22.

Exclusion Criterion:

* Has been withdrawn from the FE200486 CS14 study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2005-03; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (22):
- United States (17):
  - Urology Centers of Alabama, Homewood, Alabama
  - Advanced Urology Medical Center, Anaheim, California
  - West Coast Clinical Research, Tarzana, California
  - Western Clinical Research, Torrance, California
  - Urology Associate PC', Denver, Colorado
  - South Florida Medical Research, Aventura, Florida
  - SW Florida Urological Associates, Fort Myers, Florida
  - Northeast Indiana Research, LLC, Fort Wayne, Indiana
  - Regional Urology, Shreveport, Louisiana
  - Lawrenceville Urology, Lawrenceville, New Jersey
  - The Urology Center, Greensboro, North Carolina
  - State College Urologic Association, State College, Pennsylvania
  - University Urological Research Institute, Providence, Rhode Island
  - Urology San Antonio Research, San Antonio, Texas
  - University of Vermont, Dept of Surgery, South Burlington, Vermont
  - Virginia Urology Center, Richmond, Virginia
  - Investigational site, Seattle, Washington
- Canada (5):
  - Can-Med Clinical Research, Inc., Victoria, British Columbia
  - The Male and Female Health and Research Centers, Barrie, Ontario
  - Brantford Urology Research, Brantford, Ontario
  - Burlington Professional Care, Burlington, Ontario
  - The Female/Male Health Centres, Oakville, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed the main FE200486 CS14 study were asked to continue into the FE200486 CS14A extension study.
Pre-assignment Details: 127 participants started and 87 participants completed the main CS14 study. Of these, 57 participants were recruited into the extension study CS14A and 34 participants signed the informed consent for dose shift.
Period: Overall Study
Arm/Group | Degarelix (60 mg to 160 mg) | Degarelix (80 mg to 160 mg)
Started | 30 (Safety analysis set) | 27
Switched to Higher Dose | 17 (A protocol amendment changed the dosage to 160 mg (40 mg/mL)) | 17
Completed | 2 (Participants ongoing at the time of study closure were considered to have completed the study) | 6
Not Completed | 28 | 21
Not completed — Adverse Event | 12 | 6
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 3 | 3
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Physician Decision | 3 | 7
Not completed — Lack of Efficacy | 2 | 1
Not completed — Research site closing | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix (60 mg to 160 mg) | Degarelix (80 mg to 160 mg) | Total
Number analyzed (Participants) | 30 | 27 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] — Safety analysis set
  years | 76.0 (6.63) | 74.1 (8.85) | 75.1 (7.75)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety analysis set
  Participants
    Female | 0 | 0 | 0
    Male | 30 | 27 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants] — Safety analysis set
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 5 | 2 | 7
    White | 24 | 25 | 49
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Body weight [Mean (Standard Deviation); unit: kilogram] — Safety analysis set
  kilogram | 79.0 (11.4) | 81.3 (13.3) | 80.1 (12.2)
Body mass index [Mean (Standard Deviation); unit: kilogram per square meter] — Safety analysis set
  kilogram per square meter | 26.5 (3.64) | 26.6 (4.63) | 26.5 (4.10)
Curative Intent [Number; unit: participants] — Safety analysis set. A curative intent of Yes refers to participants who have been castrated via radical prostatectomy or radiotherapy.
  participants
    Yes | 11 | 11 | 22
    No | 19 | 16 | 35
Gleason Score [Number; unit: participants] — Safety analysis set. The Gleason score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10, with low numbers being the least aggressive and 10 being the most aggressive.
  participants
    2-4 | 2 | 1 | 3
    5-6 | 5 | 8 | 13
    7-10 | 23 | 18 | 41
Stage of Prostate Cancer [Number; unit: participants] — Safety analysis set. Prostate cancer stage was classified to describe the extent of cancer. Localized refers to tumors without involvement of lymph nodes or metastasis. Advanced localized can be larger tumors that may involve the lymph nodes but no metastasis. Metastatic are more advanced cancers that are spreading beyond the original tumor.
  participants
    Localized | 14 | 7 | 21
    Locally advanced | 3 | 5 | 8
    Metastatic | 5 | 5 | 10
    Not classifiable | 8 | 10 | 18
Time since Prostate Cancer Diagnosis [Mean (Standard Deviation); unit: days] — Safety analysis set
  days | 1253 (1565) | 1349 (1625) | 1299 (1580)

OUTCOME MEASURES:

1. Primary Outcome: Participants With Markedly Abnormal Change in Vital Signs and Body Weight
Description: This outcome measure included incidence of markedly abnormal changes in blood pressure (systolic and diastolic), pulse, and body weight at the end of trial as compared to baseline. The table presents the number of participants in each group with normal baseline and markedly abnormal value post-baseline.
Time Frame: 5 years
Population: The data include data from participants participating in both the main study (FE200486 CS14) and the extension study FE200486 CS14A.
Measure: Number; unit: participants
Arm/Group | Degarelix (60 mg to 160 mg) | Degarelix (80 mg to 160 mg)
Number analyzed (Participants) | 30 | 27
participants
  Diastolic blood pressure <=50 and decrease >=15 | 9 | 4
  Diastolic blood pressure >=105 and increase >=15 | 3 | 3
  Systolic blood pressure <=90 and decrease >=20 | 3 | 7
  Systolic blood pressure >=180 and increase >=20 | 5 | 4
  Heart rate <=50 and decrease >=15 | 2 | 6
  Heart rate >=120 and increase >=15 | 1 | 0
  Body weight decrease of >=7 percent | 6 | 4
  Body weight increase of >=7 percent | 6 | 5

2. Primary Outcome: Liver Function Tests
Description: The figures present the number of participants who had abnormal (defined as above upper limit of normal range (ULN)) alanine aminotransferase (ALT) levels, aspartate aminotransferase levels, and bilirubin levels plus the number of participants who had ALT increases >3x ULN and ALT increases >3x ULN with concurrently increased bilirubin >1.5 ULN.
Time Frame: 5 years
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Degarelix (60 mg to 160 mg) | Degarelix (80 mg to 160 mg)
Number analyzed (Participants) | 30 | 27
participants
  Abnormal alanine aminotransferase (ALAT) | 8 | 11
  Abnormal aspartate aminotransferase | 5 | 4
  Abnormal bilirubin | 7 | 5
  ALAT >3x upper limit of normal (ULN) | 0 | 0
  ALAT >3x ULN, bilirubin >1.5x ULN | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 years.
Description: Each participant's condition was monitored throughout the trial from the time of signing the informed consent until the end of the follow-up period. The investigator was to record all adverse events (AEs) in the AE log of the participant's Case Report Form.
Arm/Group | Degarelix (60 mg to 160 mg) | Degarelix (80 mg to 160 mg)
Serious Adverse Events (participants affected / at risk) | 11/30 | 7/27
Other Adverse Events (participants affected / at risk) | 29/30 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix (60 mg to 160 mg) (N=30) | Degarelix (80 mg to 160 mg) (N=27)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
General physcial health deterioration (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Appendiceal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Metastasis to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix (60 mg to 160 mg) (N=30) | Degarelix (80 mg to 160 mg) (N=27)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Atrioventricular block first degree (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Bundle branch block left (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 2 (3) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (5)
Nausea (Gastrointestinal disorders) | 5 (6) | 2 (2)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 8 (11) | 5 (9)
Injection site pain (General disorders) | 7 (18) | 6 (19)
Injection site nodule (General disorders) | 7 (16) | 5 (14)
Injection site erythema (General disorders) | 3 (18) | 5 (14)
Chills (General disorders) | 2 (4) | 5 (8)
Injection site induration (General disorders) | 1 (1) | 4 (6)
Oedema peripheral (General disorders) | 2 (2) | 2 (5)
Injection site haematoma (General disorders) | 2 (2) | 1 (4)
Injection site mass (General disorders) | 1 (6) | 2 (2)
Injection site reaction (General disorders) | 1 (1) | 2 (3)
Pain (General disorders) | 2 (3) | 1 (2)
Pyrexia (General disorders) | 1 (1) | 2 (3)
Asthenia (General disorders) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 2 (3)
Injection site warmth (General disorders) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 5 (9) | 6 (8)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 6 (7)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Tooth abscess (Infections and infestations) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 2 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Weight increased (Investigations) | 4 (4) | 7 (7)
Prostatic specific antigen increased (Investigations) | 5 (5) | 1 (1)
Weight decreased (Investigations) | 2 (3) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (3) | 1 (1)
Haemoglobin decreased (Investigations) | 3 (3) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 4 (6) | 5 (6)
Headache (Nervous system disorders) | 2 (2) | 2 (3)
Insomnia (Psychiatric disorders) | 3 (4) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 3 (3) | 3 (3)
Dysuria (Renal and urinary disorders) | 1 (1) | 4 (5)
Micturition urgency (Renal and urinary disorders) | 2 (2) | 3 (4)
Nocturia (Renal and urinary disorders) | 0 (0) | 5 (8)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 2 (3) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 2 (2) | 2 (4)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Pruritus genital (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (7) | 5 (6)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hot flush (Vascular disorders) | 12 (15) | 15 (19)
Hypertension (Vascular disorders) | 4 (4) | 4 (6)
Hypotension (Vascular disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript.